CLINICAL TRIAL: NCT01986426
Title: A Phase I, Open-label, Multi-arm, Multi-centre, Multi-dose, Dose Escalation Study of LTX-315 as Monotherapy or in Combination With Either Ipilimumab or Pembrolizumab in Patients With Transdermally Accessible Tumours
Brief Title: LTX-315 in Patients With Transdermally Accessible Tumours as Monotherapy or Combination With Ipilimumab or Pembrolizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Collaborators: Theradex (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C12-315-03
Record Dates: First submitted 2013-10-28; First posted 2013-11-18 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Melanoma; Breast Cancer; Head and Neck Cancer; Lymphoma; Triple-Negative Breast Cancer
Keywords: Transdermal accessible tumours
MeSH Terms: conditions — Neoplasms; Melanoma; Breast Neoplasms; Head and Neck Neoplasms; Lymphoma; Triple Negative Breast Neoplasms | interventions — LTX-315; Ipilimumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A: LTX-315 monotherapy singe lesion (Experimental): Cohort 1-3: First induction treatment (6 weeks): In week 1 the first index lesion will be injected Twice daily on 3 consecutive days. During week 2-6 the injection will be once a week.
  Second induction treatment (6 weeks) and Maintenance treatment (20 weeks)- At week 7 the second index lesion will be injected with same dosing schedule as the first index lesion.
  Cohort 4 and above: Once daily on 3 consecutive days week 1. Week 2-6 one injection per week. From week 8, one dosing days every 2 weeks.
  Interventions: Drug: LTX-315 consecutive lesions
- Arm B: LTX-315 monotherapy in multiple concurrent lesions (Experimental): Patients with at least one injectable lesion and one bystander lesion will receive LTX-315 to one or more lesions:
  Once daily on 2 consecutive days week 1-3.
  Interventions: Drug: LTX-315
- Arm C (Experimental): Patients with melanoma and at least one injectable lesion will receive LTX-315 to one or more lesions on two consecutive days week 1-3 in combination with ipilimumab given for 4 cycles every 3 weeks.
  Interventions: Drug: LTX-315 + ipilimumab
- Arm D (Experimental): Patients with TNBC and at least one injectable lesion will receive LTX-315 to one or more lesions on two consecutive days week 1-3 in combination with pembrolizumab given every 3 weeks.
  Interventions: Drug: LTX-315 + pembrolizumab

INTERVENTIONS:
Drug: LTX-315 consecutive lesions — Dose escalation:
  Cohort 1: 2 mg twice per day (4 mg) Cohort 2: 3 mg twice per day (6 mg) Cohort 3: 4 mg twice per day (8 mg)
  Other Names: Protocol version 4
  Arms: Arm A: LTX-315 monotherapy singe lesion
Drug: LTX-315 — Dose escalation:
  Cohort 1: 3 mg per injection Cohort 2: 4 mg per injection Cohort 3: 5 mg per injection
  Other Names: Arm B (Protocol version 6)
  Arms: Arm B: LTX-315 monotherapy in multiple concurrent lesions
Drug: LTX-315 + ipilimumab — Cohort 1: 3 mg per injection + 3 mg/kg ipilumumab Cohort 2: 4 mg per injection + 3 mg/kg ipilumumab Cohort 3: 5 mg per injection + 3 mg/kg ipilumumab
  Other Names: Arm C (Protocol version 6)
  Arms: Arm C
Drug: LTX-315 + pembrolizumab — Cohort 1: 3 mg per injection + 200 mg pembrolizumab Cohort 2: 4 mg per injection + 200 mg pembrolizumab Cohort 3: 5 mg per injection + 200 mg pembrolizumab
  Other Names: Arm D (Protocol version 6)
  Arms: Arm D

SUMMARY:
The study will assess the safety, tolerability, PK and efficacy of different intra-tumoral dosing regimens of LTX-315; a lytic-peptide that induces long-term anti-cancer immune responses, as monotherapy or in combination with ipilimumab or pembrolizumab.

DETAILED DESCRIPTION:
In this phase I, open-label, multi-arm, multicentre, multi-dose dose escalation study in patients with transdermally accessible tumours; the safety, PK and efficacy of different dosing regimens of LTX-315 will be assessed.

Patients will be allocated into 4 separate (parallel) arms depending on the tumour type and the number of lesions available.

Arm A: Single lesion/sequential lesion treatment arm (LTX-315 monotherapy) (Completed) Arm B: Concurrent multiple lesion treatment arm with all tumour types (LTX-315 monotherapy) Arm C: LTX-315 combination with ipilimumab in patients with melanoma Arm D: LTX-315 combination with pembrolizumab in patients with TNBC

All patients will have at least one lesion available for injection.

Treatment schedule:

Arm A: Injection of LTX-315 3 days week 1, 1 day in week 2, 3, 4, 5 and 6. Every 2 weeks starting with week 8.

Arm B (all tumours): Injection of LTX-315 2 days week 3 weeks (Day 1, 2, 8, 9, 15 and 16).

Arm C (melanoma): Injection of lTX-315 2 days week 3 weeks (Day 1, 2, 8, 9, 15 and 16) in combination with ipilimumab given in week 1 and every 3 weeks 4 cycles.

Arm D (TNBC): Injection of LTX-315 2 days week 3 weeks (Day 1, 2, 8, 9, 15 and 16) in combination with pembrolizumab given in week 1 and every 3 weeks up to 2 years.

Patients will be enrolled into a dose cohort in order of study entry. Staring with the lowest dose. A minimum of 3 patients will be enrolled into each cohort. Dose escalation determined by the Safety Review Committee and the Sponsor. The the optimal regimen will be based on the results of the Dose Escalation from the following information:

1. Safety parameters including blood samples and cardiovascular effects
2. Immunohistology and ultrasound confirmation of necrosis and tumour infiltrating lymphocytes
3. Systemic inflammatory response
4. Evidence of clinical responses

Cohorts may be utilized to:

1. Evaluate different doses of LTX-315
2. Explore potential modifications to the dosing schedule
3. Evaluate the potential to include appropriate combination therapies with LTX-315
4. Gain further information on clinical efficacy

ELIGIBILITY:
Inclusion Criteria:

Arm A: (Recruitment completed)

Arm B:

* Unresectable metastatic disease (any tumor type) and conventional anti-tumor treatment is not appropriate.
* Have at least one available lesion (cutaneous, sub-cutaneous, oral or lymph node) for injection between 1-3 cm longest diameter and one bystander lesion (non-injected).

Arm C:

* Have unresectable/metastatic diagnosis of malignant melanoma (histologically confirmed).
* Have at least one available lesion (cutaneous, sub-cutaneous, oral or lymph node) for injection and biopsy which is between 1 and 3 cm in longest diameter.
* Have had previous treatment with an anti-PD-1 antibody (as monotherapy or as part of combination (any combination) as 1st or 2nd line metastatic treatment).

Arm D:

* Have unresectable/metastatic diagnosis of triple negative breast cancer (histologically confirmed).
* Have at least one available lesion (cutaneous, sub-cutaneous or lymph node) for injection and biopsy with a minimum longest diameter of 1 cm.
* Have received between one and 4 prior systemic treatments for metastatic triple negative breast cancer.

All arms:

* Be willing to undergo repeat tumour biopsy and/or tumour resection procedures.
* Have an ECOG Performance status (PS): 0 - 1.
* Meet the following laboratory requirements:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  2. Absolute lymphocyte count ≥ 0.8 x 109/L
  3. Platelet count ≥ 75 x 109/L
  4. Haemoglobin ≥ 9.0 g/dL
  5. aPTT/PT within the institution's normal range
  6. Total bilirubin level ≤ 1.5 x ULN
  7. ASAT and ALAT ≤ 2.5 x ULN (≤5 x ULN if liver metastasis present)
  8. Creatinine ≤ 1.5 x ULN
  9. Albumin ≥ 30 g/L

     Exclusion Criteria:

     Arm A: (Completed)

     Arm B:
* Have a history of systemic auto-immune disease requiring anti-inflammatory or immunosuppressive therapy within the last 3 months. Patients with history of autoimmune thyroiditis are eligible provided the patient requires only thyroid hormone replacement therapy and disease has been stable for ≥ 1 year.

Arm C:

* Have had prior therapy with ipilimumab or any other anti-CTLA-4 monoclonal antibody.
* Have had BRAF/MEK inhibitors administered within 2 weeks prior to the study drug administration.
* Have active systemic autoimmune disease; have had prior pneumonitis; have a history of severe hypersensitivity to another monoclonal antibody; are receiving immunosuppressive therapy; have a history of severe immune-related adverse reaction from treatment with a monoclonal antibody, defined as any Grade 4 or 3 toxicity requiring corticosteroid treatment (> 10 mg/day prednisone or equivalent) for greater than 12 weeks.

Arm D:

* Have had prior therapy with an anti-PD-1 or anti-PD-L1 monoclonal antibody.
* Have received cancer immunotherapy within 2 weeks prior to study drug administration or have not recovered from adverse events (to ≤ CTCAE grade 1) due to such agents.
* Have active systemic autoimmune disease; have had prior pneumonitis; have a history of severe hypersensitivity to another monoclonal antibody; are receiving immunosuppressive therapy; and have a history of severe immune-related adverse reactions from treatment with a monoclonal antibody, defined as any Grade 4 or 3 toxicity requiring corticosteroid treatment (> 10 mg/day prednisone or equivalent) for greater than 12 weeks.

All arms:

* Have received external radiotherapy or cytotoxic chemotherapy within 4 weeks prior to study drug administration, or have not recovered from adverse events (≤ CTCAE grade 1) due to agents administered more than 4 weeks earlier. Palliative radiotherapy to non-target lesions within 4 weeks prior to study drug administration is allowed.
* Are currently taking any agent with a known effect on the immune system. Patients are allowed to be on a stable dose of corticosteroids (up to 10 mg daily prednisolone or equivalent) for at least 2 weeks prior to study drug administration (please see Appendix IV for prohibited medications).
* Have any other serious illness or medical condition such as, but not limited to:

  1. Uncontrolled infection or infection requiring antibiotics
  2. Uncontrolled cardiac failure: Classification III or IV (New York Heart Association)
  3. Uncontrolled systemic and gastro-intestinal inflammatory conditions
  4. Bone marrow dysplasia
* Have a known history of positive tests for HIV/AIDS, or have active hepatitis B or C (based on serology).
* Are expected to need any other anti-cancer therapy or immunotherapy to be initiated during the study period.

  15. Have clinically active or unstable CNS metastases as assessed by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 21 days
  Dose limiting toxicities (DLT) and the overall safety profile (adverse events (AE), laboratory assessments, physical findings and symptomatic assessment) of LTX-315 as monotherapy and in combination with ipilimumab or pembrolizumab.

SECONDARY OUTCOMES:
Anti tumour activity in injected tumour | Every 8 weeks from treatment start up to 24 months or first documented progression documented assessed
  Number of patients with regression of injected tumour assessed by ultrasound and/or CT/MRI.
Complete response (irCR) and partial response (irPR) | Every 8 weeks from treatment start up to 24 months or first documented progression documented assessed
  Number of patients by irRC
Overall response rate (OR) | Every 8 weeks from treatment start up to 24 months or first documented progression documented assessed
  (irRC criteria)
Disease control rate (CR + PR + SD) | Every 8 weeks from treatment start up to 24 months or first documented progression documented assessed
  irRC criteria
Progression free survival (PFS) | Every 8 weeks from treatment start up to 24 months or first documented progression documented assessed
  irRC criteria

OTHER OUTCOMES:
Pharmacokinetic (PK) profile of LTX-315 | Pre and 1 hour post dosing Day 2 Week 1
  Measurement of plasma concentrations of LTX-315 pre- and 1 hour post-dosing day 2 in week 1.

CONTACTS AND LOCATIONS:
Overall Officials: James Spicer, MD, PhD, Principal Investigator — Guy's Hospital
Locations (14):
- Belgium (2):
  - Jules Bordet Institute, Brussels
  - Cliniques Universitaires St-Luc, Service d'oncologie médicale, Brussels
- France (2):
  - Institut Curie, Paris
  - Institute Gustave Roussy, Paris
- Italy (4):
  - Intotuto Europeo di Oncologia (IEO), Milan
  - San Raffaele Hospital, Milan
  - Intituto Nazionale dei Tumori, Napoli
  - Instituto Oncologico Venneto (IOV), Padua
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital Radiumhospitalet, Oslo
- United Kingdom (4):
  - Guy's Hospital, London
  - Royal Marsden Hospital, London
  - University College of London Hospital, London
  - Christie Hospital NHS Foundatin Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spicer J, Marabelle A, Baurain JF, Jebsen NL, Jossang DE, Awada A, Kristeleit R, Loirat D, Lazaridis G, Jungels C, Brunsvig P, Nicolaisen B, Saunders A, Patel H, Galon J, Hermitte F, Camilio KA, Mauseth B, Sundvold V, Sveinbjornsson B, Rekdal O. Safety, Antitumor Activity, and T-cell Responses in a Dose-Ranging Phase I Trial of the Oncolytic Peptide LTX-315 in Patients with Solid Tumors. Clin Cancer Res. 2021 May 15;27(10):2755-2763. doi: 10.1158/1078-0432.CCR-20-3435. Epub 2021 Feb 4. PMID 33542073
- [Derived] Jebsen NL, Apelseth TO, Haugland HK, Rekdal O, Patel H, Gjertsen BT, Jossang DE. Enhanced T-lymphocyte infiltration in a desmoid tumor of the thoracic wall in a young woman treated with intratumoral injections of the oncolytic peptide LTX-315: a case report. J Med Case Rep. 2019 Jun 10;13(1):177. doi: 10.1186/s13256-019-2088-6. PMID 31177991